CLINICAL TRIAL: NCT02629393
Title: A Phase 2/3, Multicenter, Multinational, Open Label Study to Evaluate the Efficacy and Safety of ORGN001 (Formerly ALXN1101) in Neonates, Infants and Children With Molybdenum Cofactor Deficiency (MOCD) Type A
Brief Title: Study of ORGN001 (Formerly ALXN1101) in Neonates, Infants and Children With Molybdenum Cofactor Deficiency (MOCD) Type A
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Origin Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1101-MCD-202
Record Dates: First submitted 2015-12-03; First posted 2015-12-14 (Estimated); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Molybdenum Cofactor Deficiency, Type A
Keywords: Molybdenum Cofactor Deficiency (MoCD); Molybdenum Cofactor (MoCo) biosynthesis; sulfite oxidase (SO); S sulfocysteine (SSC); xanthine oxidoreductase; aldehyde oxidase
MeSH Terms: conditions — Molybdenum Cofactor Deficiency, Complementation Group A; Molybdenum cofactor deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ORGN001 (formerly ALXN1101) (Experimental)
  Interventions: Drug: ORGN001 (formerly ALXN1101)

INTERVENTIONS:
Drug: ORGN001 (formerly ALXN1101)

SUMMARY:
To evaluate the safety and efficacy of ORGN001(formerly ALXN1101) in neonate patients with MoCD Type A

ELIGIBILITY:
Patients must meet all of the following inclusion criteria to be considered for enrollment in this study:

1. Male or female neonatal patient (1 to 28 days of age [inclusive] at the time of ORGN001 administration, with day 1 of age corresponding to the day of birth) or infant (29 days to <2 years of age) or child (2 to 5 years of age [inclusive]) with MoCD Type A, previously untreated with ORGN001 or treated with ORGN001 through Compassionate Use/Individual Named Patient access
2. In neonates, diagnosis of MoCD Type A, based on:

   Prenatal genetic diagnosis, or Onset of clinical and/or laboratory signs and symptoms consistent with MoCD Type A (eg, seizures, exaggerated startle response, high-pitched cry, axial hypotonia, limb hypertonia, feeding difficulties, elevated urinary sulfite and/or SSC, elevated xanthine in urine or blood, or low or absent uric acid in the urine or blood) within the first 28 days after birth
3. In infants or children, diagnosis of MoCD Type A, based on:

   Confirmed genetic diagnosis (genetic confirmation of the diagnosis of MoCD Type A may be obtained after initiation of ORGN001 therapy in certain cases), biochemical profile, and clinical presentation consistent with MoCD Type A
4. Parent or legal guardian must have signed the informed consent form (ICF) prior to any study procedures being performed

Patients will be excluded from participating in the study if they meet any of the following criteria:

1. Diagnosis other than MoCD Type A (may be determined after the initiation of study drug)
2. Condition that is considered by the treating physician to be a contraindication to therapy, including evidence of abnormalities on brain imaging not attributable to MoCD Type A, or that might otherwise interfere with the patient's participation in the study, pose any additional risk for the patient, or confound patient assessments
3. Antenatal and/or postnatal brain imaging prior to initiation of treatment with ORGN001 that indicates cortical or subcortical cystic encephalomalacia, clinically significant intracranial hemorrhage, or other abnormalities on brain imaging determined by the treating physician to be clinically significant
4. Modified Glasgow Coma Scale (mGCS) for Infants and Children score of less than 7 for more than 24 hours (does not apply to children less than 1 day in age).

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liza Squires, M.D., Study Director — Origin Biosciences
Locations (11):
- United States (3):
  - Children's Hosptial of Michigan, Detroit, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- HaEmek Medical Center, Afula, Israel
- Stavanger Universitetssjukehus, Stavanger, Norway
- Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona, Spain
- Turkey (Türkiye) (3):
  - Hacettepe University of Medicine, Ankara
  - Gazi University, Ankara
  - Akdeniz University Medical Faculty, Antalya
- United Kingdom (2):
  - Willink Biochemical Genetics Unit, Manchester, Greater Manchester
  - Great Ormond Street Hosptial, London

REFERENCES:
- See also: FDA Drug Approval Package — https://www.accessdata.fda.gov/drugsatfda_docs/nda/2021/214018Orig1s000TOC.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Treated With ORGN001 (Formerly ALXN1101): All patients who received at least one dose of ORGN001 (formerly ALXN1101)
Period: Overall Study
Arm/Group | Patients Treated With ORGN001 (Formerly ALXN1101)
Started | 5
Completed | 2
Not Completed | 3
Not completed — MOCD Type A not genetically confirmed | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Only patients with genetically confirmed MOCD Type A are included
Arm/Group | Patients Treated With ORGN001 (Formerly ALXN1101)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: days old] | 1 [1 to 1004]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Norway | 1
  United Kingdom | 1
  Israel | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Patients with a confirmed diagnosis of MOCD Type A, treated with ORGN001 and still alive at last observation.
Time Frame: Through last observation (average of 24 months)
Measure: Count of Participants; unit: Participants
Groups:
- ORGN001 (Formerly ALXN1101): ORGN001 (formerly ALXN1101)
Arm/Group | ORGN001 (Formerly ALXN1101)
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Feeding Pattern
Description: Number of patients who can feed orally
Time Frame: At Month 12 visit
Measure: Count of Participants; unit: Participants
Groups:
- ORGN001 (Formerly ALXN1101): Patients with a confirmed diagnosis of MOCD Type A and treated with at least one dose of ORGN001 (formerly ALXN1101)
Arm/Group | ORGN001 (Formerly ALXN1101)
Number analyzed (Participants) | 3
Participants
  Oral feeding at Baseline: Able to feed orally | 2
  Oral feeding at Baseline: Not able to feed orally | 1
  Oral feeding at Month 12: Able to feed orally | 3
  Oral feeding at Month 12: Not able to feed orally | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected from Day 1 with ORGN001 treatment until study completion, up to Month 36 or study termination or completion.
Description: All-cause mortality is zero in this study because there were no deaths that occurred in patients with confirmed MOCD Type A.
  All SAE data presented.
Arm/Group | Patients Treated With ORGN001 (Formerly ALXN1101)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Treated With ORGN001 (Formerly ALXN1101) (N=5)
Apneoa (Respiratory, thoracic and mediastinal disorders) | 1
Complication associated with device (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Catheter site swelling (General disorders) | 1
Viral tonsillitis (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Viral infection (Infections and infestations) | 1
Gastrointestinal viral (Infections and infestations) | 1
Central venous catheterisation (Surgical and medical procedures) | 1
Device leakage (Product Issues) | 1
Cardiac failure (Cardiac disorders) | 1
Seizures (Nervous system disorders) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Treated With ORGN001 (Formerly ALXN1101) (N=5)
Pneumonia (Infections and infestations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Anal fissure (Gastrointestinal disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Pathogen resistance (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Pyrexia (General disorders) | 1
Catheter site infection (Infections and infestations) | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Chiari network (Congenital, familial and genetic disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Staphylococcus test positive (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Catheter site rash (General disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Otitis media acute (Infections and infestations) | 1
Catheter site erythema (General disorders) | 1
Catheter site haemorrhage (General disorders) | 1
Catheter site swelling (General disorders) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Viral infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Cardiac failure (Cardiac disorders) | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 1
Eye discharge (Eye disorders) | 1
Seizure (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Haematuria (Renal and urinary disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the small number of patients and no control, there was no SAP for this study. Results were reported by individual patient and were only descriptive. Results in tabular format are unavailable except for binary measures, such as survival and feeding ability. For more information and summary data, please refer to the referenced FDA approval package.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/Investigator shall have the right to publish or present the results of Institution's and Investigator's activities including that Study Data which was obtained or derived at Institution. Institution/Investigator agree to submit any proposed publication/presentation to Sponsor for review at least 60 days prior to submitting any such proposed publication. Within 30 days of its receipt, Sponsor shall advise if any changes are needed to protect confidentiality.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT02629393/Prot_SAP_000.pdf